CLINICAL TRIAL: NCT00088790
Title: Phase I Study to Assess the Safety and Tolerability of AZD5438 in Patients With Advanced Solid Malignancies
Brief Title: AZD5438 in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Purpose: Treatment
Other Study IDs: D0110C00005
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Neoplasms
Keywords: advanced, solid, malignancies
MeSH Terms: conditions — Neoplasms | interventions — AZD5438

INTERVENTIONS:
Drug: AZD5438

SUMMARY:
Purpose of this study is to assess the safety and tolerability of AZD5438 given orally to patients with advanced solid malignancies A review of the emerging clinical tolerability and exposure data from this study in conjunction with preclinical and the available clinical pharmacodynamic data relating to AZD5438, led to a decision by AstraZeneca that the development of AZD5438 as a potential anti-cancer agent would be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid malignancy
* Cancer refractory to standard treatments or for which no standard therapy exits

Exclusion Criteria:

* Radiotherapy within 3 weeks of the start of treatment
* Investigational product within the last 3 weeks
* Systemic cytotoxic anti-cancer therapy within the last 3 weeks
* Any significant clinical disorder that makes it undesirable for the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York